CLINICAL TRIAL: NCT06781346
Title: Analgesic Efficacy of Rhomboid Intercostal Block Compared With Thoracic Paravertebral Block in Adult Patients Undergoing Breast Cancer Surgeries: A Randomized Controlled Double-blinded Study
Brief Title: Rhomboid Intercostal Block Compared With Thoracic Paravertebral Block in Breast Cancer Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mahdy Ahmed Abd Elhady, Associate professor of anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M 729
Record Dates: First submitted 2024-12-17; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Pain, Postoperative
Keywords: Rhomboid Intercostal block; Breast surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhomboid intercostal block (Experimental): A 22G, 50mm block needle (SONOTAP,Pajunk, -Geisingen,Germany) will be inserted in the cranial to caudal direction via an in-plane approach between the medial border of the scapula between the 4th and 5th rib of the patients in the RIB group. In the ultrasound image, the trapezius muscle, rhomboid muscle, intercostal muscles,pleura, and lung were identified. Under the aseptic condition, inserted laterally in the plane of the T5 level guided by an ultrasound probe with an in plane technique.
  Interventions: Procedure: Rhomboid Intercostal Block
- Thoracic paravertebral block (Active Comparator): the transverse process and the pleura will be identified and needle will be inserted in the cranial to caudal direction till it pierces the SCTL and reaches the paravertebral space.
  Interventions: Procedure: Thoracic Paravertebral Block

INTERVENTIONS:
Procedure: Rhomboid Intercostal Block — In RI block group, A 22G, 50mm block needle (SONOTAP,Pajunk, -Geisingen,Germany) will be inserted in the cranial to caudal direction via an in-plane approach between the medial border of the scapula between the 4th and 5th rib of the patients in the RIB group. In the ultrasound image, the trapezius muscle, rhomboid muscle, intercostal muscles,pleura, and lung were identified. Under the aseptic condition, inserted laterally in the plane of the T5 level guided by an ultrasound probe with an in plane technique. The intravascular injection should be confirmed negative through aspiration, and 1-3 ml of normal saline was injected to divide the rhomboid and intercostal muscle, and a total volume of 20 ml of bupivacaine 0.25% ( not exceeding a maximum dose of 2 mg/kg) will be injected After negative aspiration of blood or air, injected into the deep layer of the rhomboid muscle.
  Arms: Rhomboid intercostal block
Procedure: Thoracic Paravertebral Block — In the TPV block group , the transverse process and the pleura will be identified and needle will be inserted in the cranial to caudal direction till it pierces the SCTL and reaches the paravertebral space. After negative aspiration of blood or air a total volume of 20 ml of bupivacaine 0.25% will be injected displacing the pleura downwards.
  Arms: Thoracic paravertebral block

SUMMARY:
Postoperative pain is a significant problem following breast surgery . If not treated in time, it may lead to delayed wound healing, respiratory depression, hemodynamic disorders, anxiety,other complications, and finally lead to difficult recovery of patients . Therefore, the prevention of postoperative pain is of great importance for patients.

Opioids, while effective in pain management, are linked to a spectrum of adverse effects, including respiratory depression, post-operative nausea and vomiting, pruritus and constipation. The adoption of multimodal analgesia following breast cancer surgery emerges as a pivotal strategy to mitigate the complications associated with opioid use in the postoperative period.[4] US-guided rhomboid intercostal block (US-RIB) is a new fascial block technique discovered by Elsharkawy et al in 2016.

Injection of local anaesthetic into the fascial plane between rhomboid major and intercostal muscles provided analgesia for both the anterior and posterior hemithorax,targets the lateral cutaneous branches of the ventral rami of the thoracic intercostal nerves from T2 to T9.

Some clinical studies have reported that RIB can effectively reduce postoperative pain, reduce opioid consumption and improve the quality of recovery in patients with breast cancer surgeries .

The ultrasound guided Thoracic paravertebral (TPV) block in the context of breast cancer surgery has been reported to decrease postoperative pain score up to 72 hours, reduce opioid consumption, improve the quality of recovery, and suppress the development or decrease the severity of chronic pain by anesthetizing the spinal nerves as they emerge from the intervertebral foramina, producing ipsilateral somatosensory, visceral and sympathetic nerve blockade. TPV block involves the injection of local anesthetic (LA) into the wedge-shaped paravertebral space deep to the superior costotransverse ligament (SCTL).

In our study investigators hypothesized that the Rhomboid Intercostal block (RIB) can provide an effective analgesia comparable with thoracic paravertebral (TPV) block without the necessity to approach the pleura and the attendant risks in adult patients undergoing Breast cancer surgeries.

DETAILED DESCRIPTION:
After approval of the local institutional ethics committee and local institutional review board. Patients who are scheduled for elective breast cancer surgeries and fulfilling the inclusion criteria in Fayoum university hospital starting from june 2024 will be enrolled in this randomized controlled study until fulfilling sample size. A detailed informed consent will be signed by the eligible participants before recruitment.

The patients will be randomized into two groups: RI block group and TPV block group in a 1:1 ratio using a computer-generated random table. The patient's assigned group information will be elicited from a sealed opaque envelope by the anesthesiologist who will perform the US-guided Rl and TPV block and will not be involved in further data collection or patient care. The patients and both the surgical and anesthesia teams, who are responsible for patient care and data collection will be blinded from the group assignments.

ANESTHETIC TECHNIQUE In this study,. All patients will be monitored using electrocardiography, pulse-oximetry, capnography,Non invasive Blood Pressure for blood pressure monitoring in the operating room.

After pre-oxygenation, general anesthesia will be induced with intravenous propofol (2 mg/kg) and fentanyl (1 μg/kg). After muscle relaxation with atracurium (0.5mg/kg), tracheal intubation will be performed by a cuffed endotracheal tube ,mechanical ventilation will be adjusted to maintain the end-tidal Carbon dioxide between 30 and 35 mmHg. Maintenance of anesthesia will be made using IV atracurium and inhalational anesthesia (isoflurane) starting at one minimal alveolar concentration (MAC) and will be adjusted to obtain an adequate level of anesthesia by titrating the concentration according to the BIS monitoring (BIS Complete Monitoring System P/N 185-0151 Covidien IIc, 15 Hampshire Street, Mansfield, MA 02048 USA) to keep the BIS value between 40 and 60.

After induction , the patient will be placed in the lateral decubitus position. The same anesthesiologist will perform the block.

In both groups, the T1-T12 thoracic spinal levels will be sonographically identified using a high frequency linear US probe (HFL_50, 15_6MHz). Then the probe will be placed vertically and nearly 3 cm lateral to the spinous process at the thoracic level T4/T5. The paraspinal muscles (erector spinae, trapezius, rhomboid), transverse processes , superior costo-transverse ligament (SCTL) and parietal pleura will be all identified under parasagittal scanning.

In RI block group, A 22 G, 50mm block needle (SONOTAP,Pajunk, -Geisingen,Germany) will be inserted in the cranial to caudal direction via an in-plane approach between the medial border of the scapula between the 4th and 5th rib of the patients in the RIB group. In the ultrasound image, the trapezius muscle, rhomboid muscle, intercostal muscles,pleura, and lung were identified. Under the aseptic condition, inserted laterally in the plane of the T5 level guided by an ultrasound probe with an in plane technique. The intravascular injection should be confirmed negative through aspiration, and 1-3 ml of normal saline was injected to divide the rhomboid and intercostal muscle, and a total volume of 20 ml of bupivacaine 0.25% ( not exceeding a maximum dose of 2 mg/kg) will be injected After negative aspiration of blood or air, injected into the deep layer of the rhomboid muscle.

In the TPV block group , the transverse process and the pleura will be identified and needle will be inserted in the cranial to caudal direction till it pierces the SCTL and reaches the paravertebral space. After negative aspiration of blood or air a total volume of 20 ml of bupivacaine 0.25% will be injected displacing the pleura downwards.

After 15 min , an incision will be made to perform the surgical procedure. . Continuous hemodynamic monitoring of blood pressure and heart rate will be done . If the systolic blood pressure decreased to a 20% below the baseline, 5 mg of ephedrine will be injected IV. Moreover, if the heart rate reduced to a 50 beat per minute or less , 0.5 mg of atropine will be injected IV.

Intraoperative if blood pressure increases over 20% of baseline and BIS value is between 40-60 we will give fentanyl (1 μg/kg)

At the end of the surgery, isoflurane will be discontinued and the muscle relaxant will be antagonized with neostigmine (0.04-0.08 mg/kg) and atropine (0.01 mg/kg) and will be extubated when the patient meets the following criteria: awake or arousable, hemodynamically stable, no ongoing active bleeding and warm extremities , after the return of spontaneous respiration.

At post anesthesia care unit all patients will be monitored blood pressure , heart rate and oxygen saturation , The patient's pain will be evaluated using a Visual Analog Scale (VAS) Both during rest and with cough (0: no pain, 10: worst pain ever) at time zero (postoperative when patient is fully conscious and can assess and evaluate pain) if there is pain patient will receive ketorolac 30mg IV and Paracetamol 1 gm IV

After admission at ward at the end of surgery, all patients will receive IV fentanyl via patient controlled analgesia (PCA) with concentration 10 μg/ml , with bolus 15 μg and lockout interval 10 minutes and maximum dose of 90 μg/hr with no background dose for 24 hours. Paracetamol 1 gm IV will be given every 8 hours.. The patient's pain will be evaluated using a Visual Analog Scale (VAS) (0: no pain, 10: worst pain ever) at time intervals: Time zero (when patient is fully conscious and can assess and evaluate the pain) then 30 minutes, 1 hour, 3 hours, 6 hours, 12 hours, and 24h postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older .
* American Society of Anesthesiologists (ASA) II-lll Scheduled for elective breast surgery for modified radical mastectomy, simple mastectomy, breast conservative surgery.

Exclusion Criteria:

* Patient refusal.
* Significant renal, hepatic and cardiovascular diseases.
* History of allergy to one of the study drugs.
* Any contraindication to regional anesthesia such as local infection or bleeding disorders.
* Chronic opioid use, history of chronic pain and cognitive disorders.
* Emergent surgeries

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
The total postoperative fentanyl consumption in the first 24 hours. (μg) | in the first 24 hours.
  The total postoperative fentanyl consumption in the first 24 hours. (μg)

SECONDARY OUTCOMES:
Total intraoperative fentanyl | Intraoperative
  Total intraoperative fentanyl
Blood pressure | 24 hours postoperative
  Blood pressure intraoperative
Time to first analgesic request | 24 hours postoperative
  Postoperative
VAS score | 24 hours postoperative
  Both during rest and with cough (score 0 =no pain and 10 =worst pain ever) in the two groups of the study
Complications related to the block : pleural puncture , vascular puncture and local anesthesia systemic toxicity. | Intraoperative
  Intraoperative
Complications related to IV opioids | 24 hours postoperative
  nausea and vomiting (0 = no symptoms, 1 = only nausea, 2 = nausea and vomiting), respiratory depression (respiratory rate less than 10), sedation (0 = awake and alert, 1 = quietly awake, 2 = asleep but easily arousable, 3 = deep sleep, responding to painful stimulus), pruritus(0=no symptoms, 1=mild pruritus, 2 moderate pruritus, 3 sever pruritus)
Hospital length of stay | 24 hours Postoperative
  Postoperative
Participant satisfaction will be assessed on a 4-point scale (1:excellent , 2: good 3: fair, 4: poor). | 24 hours postoperative
  Postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mahdy A Abd El-hady, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum university Hospital, El Fayoum Qesm, Faiyum Gove, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsharkawy H, Saifullah T, Kolli S, Drake R. Rhomboid intercostal block. Anaesthesia. 2016 Jul;71(7):856-7. doi: 10.1111/anae.13498. No abstract available. PMID 27291611
- [Background] Tulgar S, Selvi O, Thomas DT, Manukyan M, Ozer Z. Rhomboid intercostal block in a modified radical mastectomy and axillary curettage patient; A new indication for novel interfascial block. J Clin Anesth. 2019 May;54:158-159. doi: 10.1016/j.jclinane.2018.12.006. Epub 2018 Dec 13. No abstract available. PMID 30553225
- [Background] Piraccini E, Biondi G, Corso RM, Maitan S. The use of rhomboid intercostal block, parasternal block and erector spinae plane block for breast surgery. J Clin Anesth. 2020 Feb;59:10. doi: 10.1016/j.jclinane.2019.06.004. Epub 2019 Jun 6. No abstract available. PMID 31176954
- [Background] Tulgar S, Kiziltunc B, Thomas DT, Manukyan MN, Ozer Z. The combination of modified pectoral nerves block and rhomboid intercostal block provides surgical anesthesia in breast surgery. J Clin Anesth. 2019 Dec;58:44. doi: 10.1016/j.jclinane.2019.04.040. Epub 2019 May 7. No abstract available. PMID 31075623
- [Background] Terkawi AS, Tsang S, Sessler DI, Terkawi RS, Nunemaker MS, Durieux ME, Shilling A. Improving Analgesic Efficacy and Safety of Thoracic Paravertebral Block for Breast Surgery: A Mixed-Effects Meta-Analysis. Pain Physician. 2015 Sep-Oct;18(5):E757-80. PMID 26431130